CLINICAL TRIAL: NCT00604864
Title: Anti TNFa Treatment for Deep Endometriosis Associated Pain : a Randomised Placebo Controlled Trial.
Brief Title: Effect of Anti TNFa Upon Deep Endometriosis Associated Pain
Acronym: Infliximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Koninckx Philippe, UZ Gasthuisberg, Catholic University Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: trial_EU-0053/endometriosis
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Endometriosis
Keywords: deep endometriosis; pelvic pain; infliximab; anti TNFa
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): women with a deep endometriosis nodule of at least 1 cm in diameter; and severe pain (at least one severe pain score on Biberoglu Behrman scale)
  Interventions: Drug: anti TNFa monoclonal antibody - Infliximab
- 2 (Placebo Comparator): women with a deep endometriosis nodule of at least 1 cm in diameter; and severe pain (at least one severe pain score on Biberoglu Behrman scale)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: anti TNFa monoclonal antibody - Infliximab — Chimeric A2 (infliximab, RemicadeTM) IgG ; 100 mg infliximab IgG, Infliximab was freshly prepared immediately before each administration. Infliximab or placebo was administered as a slow infusion of 250mL on weeks 0, 2 and 6. Women were closely observed during, and for 1 hour after, the infusion in the event of any serious adverse reactions.
  Arms: 1
Drug: placebo — Placebo
  Arms: 2

SUMMARY:
Deep endometriosis associated pain is believed to be caused by inflammation. Anti TNFa has been proved to be an effective treatment for other inflammation related conditions as Crohn's disease Endometriosis is associated with an inflammatory response in the pelvis, which is mediated by a number of cytokines including TNF-α. It has therefore been suggested that infliximab, an anti-TNF-α monoclonal antibody, might relieve pain in affected women.

DETAILED DESCRIPTION:
In this pilot study, 21 women with severe endometriosis-associated pain and a rectovaginal nodule, at least 1 cm in diameter on clinical examination, were randomised in a 2 to 1 ratio to receive intravenous infliximab (n=14) or placebo (n=7) in the three months prior to laparoscopic laser excision of the nodule.

After a 1 month observation period, all women received three infusions of infliximab (5mg/kg) or placebo over the course of 6 weeks. Surgery was performed 3 months later and follow-up continued for a further 6 months. The primary endpoint was the total pain burden (dysmenorrhoea, deep dyspareunia and non-menstrual pain) rated on a daily basis by the patient using standard pain scales and analgesic intake as the outcome measures . Secondary endpoints included the volume of the endometriotic nodule assessed clinically and on transvaginal ultrasound, the amount of pelvic tenderness on clinical examination and the presence of other endometriotic lesions at laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* The patients (aged 18-50 years) were all recruited from a single, tertiary referral hospital at Leuven University, Belgium, specialising in the surgical treatment of severe endometriosis.
* All the women were symptomatic and scheduled for surgical excision of a rectovaginal nodule, at least 1 cm in diameter, diagnosed on the basis of clinical examination at the time of menstruation.
* All the women had a menstrual cycle occurring every 25 to 40 days.
* If previously treated with hormonal medication for endometriosis, at least 3 months must have elapsed and they must have had at least two menstrual cycles since stopping treatment.
* Unless the women had previously been sterilised, they had to agree to use a double-barrier method of contraception for the duration of the study and for up to 6 months after receiving the last infusion.
* The study was approved by the Institutional Review Board of Leuven University.
* Written, informed consent was obtained before any study related procedures were performed.

Exclusion Criteria:

* Evidence on chest x-ray in the previous 3 months of old or currently active TB, or other history/evidence of active TB, even if adequately treated
* Evidence of serious infections (such as pneumonia or pyelonephritis) in the previous 3 months
* Evidence of a documented HIV infection, active hepatitis-B or C, or an opportunistic infection (e.g. herpes zoster, cytomegalovirus, pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) in the previous 6 months
* Previous transplant surgery, a lymphoproliferative disorder or other malignancy
* Positive cervical cytology in the previous 6 months
* Previous treatment with infliximab, any drug known to affect TNF-α levels, e.g. pentoxifylline, thalidomide and etanercept, or any human/murine recombinant products
* Known allergy to murine products
* Use of other investigational drugs within 1 month of recruitment or within 5 half-lives of the investigational agent, whichever was longer
* Any haematological or biochemical abnormalities on routine screening.
* Subjects were also excluded if there was any pelvic pathology on transvaginal ultrasound scan (TVS) other than small uterine fibroids (< 4 cm in diameter) and an ovarian endometrioma or endometriotic nodule.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-02; Primary Completion 2005-02 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Endometriosis associated pain | By the clinician after 1, 2 and 3 months ; by the patient daily for 3 months

SECONDARY OUTCOMES:
decrease in volume of deep endometriosis nodule | after 1, 2 and 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philippe R Koninckx, MD, PhD, Principal Investigator — Catholic University Leuven
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] Anaf V, Simon P, El Nakadi I, Fayt I, Buxant F, Simonart T, Peny MO, Noel JC. Relationship between endometriotic foci and nerves in rectovaginal endometriotic nodules. Hum Reprod. 2000 Aug;15(8):1744-50. doi: 10.1093/humrep/15.8.1744. PMID 10920097
- [Background] Colombel JF, Loftus EV Jr, Tremaine WJ, Pemberton JH, Wolff BG, Young-Fadok T, Harmsen WS, Schleck CD, Sandborn WJ. Early postoperative complications are not increased in patients with Crohn's disease treated perioperatively with infliximab or immunosuppressive therapy. Am J Gastroenterol. 2004 May;99(5):878-83. doi: 10.1111/j.1572-0241.2004.04148.x. PMID 15128354
- [Background] D'Antonio M, Martelli F, Peano S, Papoian R, Borrelli F. Ability of recombinant human TNF binding protein-1 (r-hTBP-1) to inhibit the development of experimentally-induced endometriosis in rats. J Reprod Immunol. 2000 Oct-Nov;48(2):81-98. doi: 10.1016/s0165-0378(00)00073-5. PMID 11011074
- [Derived] Koninckx PR, Craessaerts M, Timmerman D, Cornillie F, Kennedy S. Anti-TNF-alpha treatment for deep endometriosis-associated pain: a randomized placebo-controlled trial. Hum Reprod. 2008 Sep;23(9):2017-23. doi: 10.1093/humrep/den177. Epub 2008 Jun 12. PMID 18556683